CLINICAL TRIAL: NCT03919097
Title: Retrospective Study to Identify Risk Factors for Atrial Fibrillation After Ablation of Atrial Flutter by Radiofrequency of the Cavotricuspid Isthmus.
Brief Title: Identification of Risk Factors for Atrial Fibrillation After Ablation of an Atrial Flutter by Radiofrequency of the Cavotricuspid Isthmus.
Status: Completed | Type: Observational
Sponsor: José Castro (Other)
Responsible Party: Sponsor-Investigator, José Castro, Head of cardiology clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Fayad
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: No atrial arrhythmia post-ablation of a flutter by radiofrequency of the isthmus of the cavotricuspid valva.
  Interventions: Other: Medical Data extraction
- Atrial fibrillation post ablation: Atrial arrhythmia (Atrial Fibrillation) post-ablation of a flutter by radiofrequency of the isthmus of the cavotricuspid valva.
  Interventions: Other: Medical Data extraction
- Flutter recidive: Recidive of the flutter after ablation.
  Interventions: Other: Medical Data extraction
- Atrial Fibrillation antecedents: Patients with atrial fibrillation after flutter ablation, with previous antecedents of atrial fibrillation.
  Interventions: Other: Medical Data extraction
- No Atrial Fibrillation antecedents: Patients with atrial fibrillation after flutter ablation, without antecedents of atrial fibrillation.
  Interventions: Other: Medical Data extraction

INTERVENTIONS:
Other: Medical Data extraction — Data extraction from the patient's Medical Files

SUMMARY:
Atrial flutter is a common condition that is effectively treated by ablation using radiofrequency. Due to its feasibility, effectiveness and low procedural risk, radiofrequency ablation is a first-line treatment of atrial flutter.

Several studies have been published concerning the factors associated with the occurrence of atrial fibrillation during or after flutter ablation, in patients with and without clinical history of atrial fibrillation. 26 to 46% of patients are likely to develop it, according to ECG or Holter diagnoses. The figure rises to more than 50% with a diagnosis with an implantable loop recorder.

In patients without a prior history of atrial fibrillation before ablation, anticoagulants are routinely administered 4-6 weeks after flutter removal by most cardiologists.

Although there are no specific guidelines for anticoagulation after flutter ablation, it is currently recommended to treat the patient as for atrial fibrillation. It is therefore crucial to identify in advance patients at high risk of atrial fibrillation after flutter ablation, in order to assess the appropriateness of maintaining oral anticoagulant therapy.

The objectives of this study are:

* to evaluate the frequency and identify the factors predicting the occurrence of atrial fibrillation after flutter ablation
* to determine the risk of a stroke occurring in patients with atrial fibrillation after flutter ablation.

The database consists in patients of the CHU Brugmann Hospital treated between 1996 and 2018.

ELIGIBILITY:
Inclusion Criteria:

Patients treated at the CHU Brugmann Hospital for flutter ablation by radiofrequency between 1996 and 2018.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the CHU Brugmann Hospital for flutter ablation by radiofrequency between 1996 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Age at ablation | One day
  Age of the patient at the date of the flutter ablation
Gender | One day
  Gender of the patient at the date of the flutter ablation
Antecedents of ischemic cardiomyopathy | One day
  Antecedents of ischemic cardiomyopathy (yes/no) at the date of flutter ablation
Antecedents of cardiomyopathy | One day
  Antecedents of cardiomyopathy (yes/no) at the date of flutter ablation
Antecedents of dilated cardiomyopathy | One day
  Antecedents of dilated cardiomyopathy (yes/no) at the date of flutter ablation
Diabetes | One day
  Diabetes diagnosis (yes/no) at the date of flutter ablation
Chronic pulmonal disease | One day
  Chronic pulmonal disease diagnosed at the date of flutter ablation
Cardiac surgery antecedents | One day
  Presence of cardiac surgery antecedents at the date of flutter ablation
Atrial fibrillation antecedents | One day
  Antecedents of Atrial fibrillation at the date of flutter ablation
Beta-blockers post-ablation | One day
  Prescription of Beta-Blockers after the flutter ablation (yes/no)
Amiodarone post-ablation | One year
  Prescription of amiodarone after the flutter ablation (yes/no)
Class I antiarrhythmic drugs post-ablation | One year
  Prescription of Class I antiarrhythmic drugs post-ablation
Arterial hypertension | One day
  Presence of arterial hypertension on the day of flutter ablation
Antecedents of stroke | One day
  Antecedents of stroke
Stroke after flutter ablation | One year
  Occurence of stroke after the flutter ablation
Antecedents of peripheric thromboembolic events | One day
  Antecedents of thromboembolic events on the day of flutter ablation
Peripheric thromboembolic events after flutter ablation | One year
  Thromboembolic events after flutter ablation
Atrial Fibrillation apparition delay | Up to one year
  Delay of apparition of atrial fibrillation after flutter removal
Left ventricular ejection fraction of the heart | One day
  Left ventricular ejection fraction of the heart at the day of flutter removal (echographic data)
Left atrium size of the heart | One day
  Left atrium size of the heart at the day of flutter removal (echographic data)
Pulmonary arterial pressure | One day
  Pulmonary arterial pressure at the day of flutter removal (echographic data)

CONTACTS AND LOCATIONS:
Overall Officials: Georges Fayad, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No